CLINICAL TRIAL: NCT05639699
Title: The Effect of Motivational Interviewing on the Level of Self-Efficacy and Addiction in Smoking Cessation in Nursing Students: A Single-Blind Randomized Controlled Study
Brief Title: The Effect of Motivational Interviewing on the Level of Self-Efficacy and Addiction in Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Associate Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ordu123
Record Dates: First submitted 2022-10-14; First posted 2022-12-06 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Quit Smoking
Keywords: Motivational interview; Smoking cessation; Self-efficacy; Level of addiction; Nursing students
MeSH Terms: conditions — Smoking Cessation | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Motivational interview will be done to the experimental group
  Interventions: Other: motivational interview
- I Control group (No Intervention): No intervention will be applied to the control group
- II Control group (No Intervention): No intervention will be applied to the control group

INTERVENTIONS:
Other: motivational interview — Quitting smoking with motivational interviewing
  Arms: Experimental group

SUMMARY:
This study will be carried out to determine the effect of motivational interviewing on the level of self-efficacy and addiction in smoking cessation in nursing students.

DETAILED DESCRIPTION:
This study will be carried out to determine the effect of motivational interviewing on the level of self-efficacy and addiction in smoking cessation in nursing students. The study was planned as a single-blind randomized controlled experimental study. The population of the research will be composed of students studying in the 1st, 2nd and 3rd years of Ordu University and Giresun University Faculty of Health Sciences Nursing Department and who meet the research criteria, and the sample will be 90 students determined by power analysis. In the study, 30 students from Ordu University Faculty of Health Sciences Nursing Department will be in the experimental group and 30 students in the I. control group. 30 students from Giresun University Faculty of Health Sciences Nursing Department will be in the second control group. Students in the experimental group will be given a motivational interview on quitting smoking for 40-50 minutes on average once a month for 6 months. No intervention will be applied to the students in the control groups during the research process, but a motivational interview will be applied once at the end of the research in terms of ethics. The data of the research will be collected with Personal Information Form, Fagerström Nicotine Addiction Test, Self-Efficacy Scale and Stage of Change Evaluation Form. In the study, repeated measurements will be made in the 1st month, 3rd month and 6th month. Necessary institutional permission and ethics committee approval will be obtained for the research. The analysis of the data will be done by an expert statistician in a computer environment.

ELIGIBILITY:
Inclusion Criteria:

* Being a 1st, 2nd, and 3rd year student of the Nursing Department,
* Continuing active education and training,
* Smoker at least one cigarette a day,
* Open to communication and cooperation, and
* Students who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Fourth grade,
* Having a serious psychiatric diagnosis (schizophrenia, bipolar disorder, psychotic disorder, etc.),
* Receiving professional support for smoking cessation,
* Changing schools during the research process and
* Students who do not want to continue the research will be excluded from the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy Scale | 1st, 3rd, and 6th months
  The scale was developed by Nicki, Remington and MacDonald in 1984. This scale, which was developed based on social learning theories, is related to the individual's belief that he or she can perform a desired behavior. This scale is used in smoking cessation studies. The scale was adapted to Turkish by Karancı. The scale consists of 25 questions, each of which consists of 5 items, and is likert type. Each item score in the scale ranges from 1 to 5. The individual rates the smoking status for each item in five categories ranging from "Not at all sure:1" to "Absolutely sure:5". The scores to be taken from the scale vary between 5-25, and as the score increases, the belief that one can quit smoking increases.
Fagerström Test for Nicotine Dependence | 1st, 3rd, and 6th months
  Dr. The test developed by Karl Fagerström in 1978 to evaluate the level of addiction to nicotine; It was reconsidered by Fagerström, Heatherton and Kazlowki and the Fagerström Test for Nicotine Dependence was created. In Turkish Uysal et al. Adapted by in 2004. In the test, which consists of 6 questions in total, each question is given a different score. The scale consists of 6 questions and each item is scored as 0,1,2,3, and one of the answer options should be marked. 2nd, 3rd, 5th of the scale. Since the 6th and 6th questions are 0-1 points, the points that can be obtained from the scale range from 0-10. The highest score "10" indicates the highest degree of nicotine addiction, and the lowest score "0" indicates no nicotine addiction. According to the total scores obtained as a result of the test, it is defined as 0-2: very little dependence, 3-4: little dependence, 5: moderately dependent, 6-7: high dependence, and 8-10: very high dependence.

SECONDARY OUTCOMES:
quit smoking | 1st, 3rd, and 6th months
  quit smoking

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildiz Ozdemir A, Gok Ugur H. The Effect of Motivational Interviewing on the Level of Self-Efficacy and Addiction in Smoking Cessation in Nursing Students: A Single-Blind Randomized Controlled Study. Int J Nurs Pract. 2025 Apr;31(2):e70009. doi: 10.1111/ijn.70009. PMID 40109145